CLINICAL TRIAL: NCT04715126
Title: A Randomized, Placebo-controlled, Blinded Study to Evaluate Efficacy of Oxyjun on Cardiovascular Health in Healthy Individuals.
Brief Title: Evaluate Efficacy of Oxyjun on Cardiovascular Health in Healthy Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EB/200401/OXYJUN/AH
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxyjun (Extract of Terminilia Arjuna). (Active Comparator)
  Interventions: Other: Oxyjun
- Placebo (Microcrystalline cellulose) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Oxyjun — One capsule to be taken after breakfast with water.
  Arms: Oxyjun (Extract of Terminilia Arjuna).
Other: Placebo — One capsule to be taken after breakfast with water.
  Arms: Placebo (Microcrystalline cellulose)

SUMMARY:
Terminalia arjuna, commonly known as arjuna, that belongs to the family of Combretaceae. Most clinical and experimental studies for Terminalia arjuna, have suggested that the crude drug possesses anti-ischemic, antioxidant, hypolipidemic, and antiatherogenic activities.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant of either sex, aged ≥ 30 to ≤ 70 years at the time of screening (completed). 2. Participants with normal to high normal blood pressure (BP) [systolic BP ≥ 120 and ≤ 139 mm Hg and/or diastolic BP ≥ 80 and ≤ 89 mm Hg] as defined by "The Task Force for the management of arterial hypertension of the European Society of Cardiology (ESC) and the European Society of Hypertension (ESH)". 3. Participants with normal to mildly deranged 'Left ventricular ejection' as per as per American College of Cardiology: LVEF ≥ 39 and ≤ 55%. 4. BMI ≥ 25 to ≤ 34.9 kg/m2 5. Normal level of Aspartate transaminase (AST) and Alanine transaminase (ALT) as specified by reference range of College of American Pathologists certified laboratory. 6. Normal level of Creatinine as specified by reference range of College of American Pathologists certified laboratory. 7. Participants must have demonstrated their willingness to participate in the study and comply with the study procedures and required visits. 8. Willing to abstain from caffeine, alcohol and related products consumption 12 hours prior to study visits. 9. Those having the ability to understand and sign a written informed consent form, which must be completed prior to study specific requirements being performed. 10. Must be literate and have the ability to complete the study-based questionnaires and requirements. 11. Female participants of childbearing age must be willing to use the accepted methods of contraception during the study.

Exclusion Criteria:

* Systolic BP ≥140 mm Hg and/ or Diastolic BP ≥ 90 mm Hg. 2. Fasting blood sugar ≥ 126 mg/dL 3. Presence of any unstable, acutely symptomatic, or life-limiting illness. 4. History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic or neurologic disorders that, in the judgment of the investigator, would interfere with the participant's ability to provide informed consent, comply with the study protocol (that might confound the interpretation of the study results), or put the participant at undue risk. 5. Using Omega fish oil supplements, anticonvulsants, Coenzyme Q10, Vitamin K2, proton pump inhibitors, loop diuretics, anticoagulants, barbiturates, anti-epileptic medications and any herbal supplements (e.g. flax seeds, chia seeds). 6. Chronic use of anti-inflammatory medications (≥ 5 tablets/20 days in last 3 months). 7. Individuals having a history of smoking or currently smoking and also using any form of smokeless tobacco. 8. High-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week for women and 5 or more alcohol containing beverages on any day or 15 or more alcohol containing beverages per week for men. 9. Binge drinkers as defined by consumption of 4 or more alcohol containing beverages for women and 5 or more alcohol containing beverages for men within 2 hours. 10. Abnormal thyroid stimulating hormone (TSH) levels beyond the defined reference range (<0.4 and > 4.0 IU/ml) 11. Participants unable to walk. 12. Participants with history of chronic caffeine use. 13. Participants who have any other disease or condition, or are using any medication, that in the judgment of the investigator would put him/her at unacceptable risk for participation in the study or may interfere with evaluations in the study or noncompliance with treatment or visits. 14. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives. 15. Females undergoing hormone replacement treatments. 16. Menopausal females having less than 3 years of menopausal history 17. Those unwilling to abstain from other dietary supplements or medication (e.g. Hepatoprotective agents and other traditional medicines - Ayurveda, Siddhi, Chinese herbal medicine, Naturopathy). 18. Have participated in a study of an investigational product 90 days prior to the screening. 19. Participants with known or suspected hypersensitivity or intolerance to Investigational product. 20. Participants who are unable to comply with study requirements. 21. Any clinical signs or symptoms that in the opinion of investigator, can jeopardize the outcome of the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Left ventricle ejection fraction | Day 0 to Day 56
  1. To evaluate the effect of 8-week consumption of Oxyjun on cardiac pumping capacity of study participants as evaluated by Left ventricle ejection fraction (LVEF).

SECONDARY OUTCOMES:
Early filling (E) and the atrial phase (A) will be calculated at rest and the E/A ratio | Day 0 to Day 56
  Reduction in myocardial stress of study participants as evaluated by decrease in E/A ratio at the end of week 8 (day 56) from baseline as compared to placebo.
Myocardial stress | Day 0 to Day 56
  Decline in myocardial stress of study participants as assessed by decrease in rate pressure product at the end of week 8 (day 56) from baseline (day 0) as compared to placebo.
Fatigue severity scale | Day 0, Day 28, day 56
  Reduction in fatigue of study participants as assessed by decrease in Fatigue severity scale at week 4 (day 28), and week 8 (day 56) from baseline (day 0) as compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanjay Wani, BAMS, Principal Investigator — Shop No.1,VardhmanApartment, Lokmanya Tilak Road,Dahisar west, Mumbai-400068.
Locations (4):
- India (4):
  - Dr. Awate clinic, Mumbai, Maharashtra
  - Shree Polyclinic,, Mumbai, Maharashtra
  - Dr Rajesh Kewalramani Clinic, Mumbai, Maharashtra
  - Dr. Wani's Clinic, Mumbai, Maharashtra